CLINICAL TRIAL: NCT04160884
Title: Fluorescence-navigated Thoracoscopy for Pulmonary Segmentectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Collaborators: Beijing Municipal Science & Technology Commission (Other)
Responsible Party: Principal Investigator, Jun Wang, Chief，Thoracic Surgery Service, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018PHB143-01
Record Dates: First submitted 2019-11-10; First posted 2019-11-13 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Pulmonary Segmentectomy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A (Active Comparator): 0.6mg/kg of ICG, iv
  Interventions: Procedure: Indocyanine Green Injection through Peripheral Vein
- B (Experimental): 0.2mg/kg of ICG, iv
  Interventions: Procedure: Indocyanine Green Injection through Peripheral Vein

INTERVENTIONS:
Procedure: Indocyanine Green Injection through Peripheral Vein — After ligation of the segmental pulmonary artery supplying the targeted segment, indocyanine is injected intravenously at a specific concentration intraoperatively.

SUMMARY:
Recently developed fluorescence-navigated thoracoscopy with indocyanine green (ICG) is being used for various kinds of pulmonary surgery, and several studies have reported the application of this novel technique in demarcation of the intersegmental border for segmentectomy. This study is performed prospectively to find out, for the first time, the optimal dosage of ICG in human body to ensure safe and sustained imaging during segmentectomy.

ELIGIBILITY:
Inclusion Criteria:

* Suitable for segmentectomy and signed informed consent

Exclusion Criteria:

* Liver dysfunction.
* Allergic to indocyanine green.
* Can't tolerate thoracoscopic surgery.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2018-12-12 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Signal-to-background Ratio (SBR) of the Targeted and Non-targeted Segments | Surgery
  We use image analysis software ImageJ to evaluate the strength of luminosity in the targeted and non-target segments using intraoperative images and calculate signal-to-background-ratio.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China